CLINICAL TRIAL: NCT05522075
Title: Reducing Blood Pressure in Mid-life Adult Binge Drinkers: the Role of Microvascular Function and Sympathetic Activity
Brief Title: Reducing Blood Pressure in Mid-life Adult Binge Drinkers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2200-0189; 4R00AA028537-03 (NIH)
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-01

CONDITIONS: Alcohol Drinking; Binge Drinking; Blood Pressure; Alcohol Abstinence; Aging; Lifestyle Factors; Vasodilation; Behavioral Problem
Keywords: Exercise training; High-intensity interval training; Midlife adults; Middle-aged; Microvascular function; Sympathetic nerve activity
MeSH Terms: conditions — Alcohol Drinking; Binge Drinking; Alcohol Abstinence; Aneurysm; Problem Behavior | interventions — Exercise; Ethanol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise Group (Experimental): Binge drinkers who have been assigned to exercise group will receive baseline assessment, 8-week exercise training plus alcohol abstinence intervention, and post-intervention assessment.
  Interventions: Behavioral: Exercise Training; Behavioral: Alcohol Abstinence Intervention
- Non-exercise Group (Active Comparator): Binge drinkers who have been assigned to non-exercise group will receive baseline assessment, 8-week alcohol abstinence intervention, and post-intervention assessment.
  Interventions: Behavioral: Alcohol Abstinence Intervention
- Alcohol abstainer/moderate drinker group (No Intervention): Alcohol abstainer/moderate drinker will complete baseline assessment only and will not receive any intervention.

INTERVENTIONS:
Behavioral: Exercise Training — Subjects will be asked to perform exercise training (high-intensity interval training) under supervision, 3 times per week for 8 weeks. Each training session will last 40 minutes and will consist of 10-minute warm up at 70% of maximal heart rate (HRmax), four 4-minute intervals at 90% of HRmax with 3-min active recovery at 70% of HRmax and 5-minute cool down at 70% of HRmax.
  Arms: Exercise Group
Behavioral: Alcohol Abstinence Intervention — Subjects will be asked to abstain from alcohol for 8 weeks. Education materials and bi-weekly consultations will be provided.
  Arms: Exercise Group; Non-exercise Group

SUMMARY:
This study has two phases:

Phase 1 is to examine blood pressure, microvascular function, and sympathetic nerve activity in mid-life adult binge drinkers vs. alcohol abstainers/moderate drinkers.

Phase 2 is to examine the effect of 8-week aerobic exercise training on blood pressure, microvascular function, and sympathetic nerve activity in mid-life adult binge drinkers

DETAILED DESCRIPTION:
During phase 1, we will measure blood pressure, microvascular function, and sympathetic nerve activity (baseline assessment) in mid-life adult binge drinkers, alcohol abstainers, and moderate drinkers. Only mid-life adult binge drinkers will enter Phase 2 and be randomized to the exercise training group and non-exercise control group. After 8 weeks of intervention, we will re-measure blood pressure, microvascular function, and sympathetic nerve activity (post-intervention assessment) in mid-life adult binge drinkers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (50-64 years of age) who do not drink alcohol, who drink at moderate levels, or who binge drink
* Female subjects will be postmenopausal (i.e., cessation of menses for ≥1 yr).
* Subjects who can speak and understand English.

Exclusion Criteria:

* a history of diabetes, cardiovascular disease, liver, or renal disease
* current or history of smoking and illicit drug use
* blood pressure ≥160/100 mm Hg
* other known traditional cardiovascular disease risks: obesity (BMI≥35 kg/m2), or hyperlipidemia (total cholesterol>230 mg/dl and/or LDL cholesterol>160 mg/dl)
* active infection (in the past 2 months)
* a history of seizures, cancer, or inflammatory disease (i.e., gout or rheumatoid)
* unstable body weight (>5% change during the past 6 months)
* regular aerobic exercise training (i.e., they engage in 30 min of structured aerobic exercise at least 3 times per week)
* current use of hormone replacement therapy (i.e., estrogen, progesterone, and testosterone)

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of high-intensity interval training | Through out the study participation (~3 months)
  Recruitment capacity (e.g., how many subjects respond and enter to the study or reasons of refusal), resulting subject characteristics, the number of exercise session attended, and the number of dropouts

SECONDARY OUTCOMES:
Changes in microvascular function | Baseline and after an 8-week intervention
  A small amount of fat will be taken form the buttock. Small vessels will then be found in the fat and their sizes in response to various flows and chemical agents will be measured.
Changes in sympathetic activity | Baseline and after an 8-week intervention
  A small electrode will be inserted into the back of the knee to record nerve activity (bursts/min).
Changes in urine catecholamine levels | Baseline and after an 8-week intervention
  Urine samples will be collected for 24 hours to measure norepinephrine levels (ug/g)
Changes in blood pressure | Baseline and after an 8-week intervention
  Systolic and Diastolic blood pressure will be measured at rest and for 24 hours.
Changes in alcohol intake | Baseline and after an 8-week intervention
  Questionnaires will be used to determine alcohol intake.

CONTACTS AND LOCATIONS:
Overall Officials: Chueh-Lung Hwang, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will submit to the NIMH Data Archive human subjects' data that were collected as part of the "Research Project" including microvascular function, sympathetic activity, and blood pressure. These data will be made accessible to authorized users for the purpose of scientific investigation, scholarship or teaching, or other forms of research and research development.
Time Frame: Data will be shared with authorized users upon publication (via an NDA Study) or 1-2 years after the grant end date (04/30/2026).
Access Criteria: Submit a Data Access Request to NDA and get approval
URL: https://nda.nih.gov/get/access-data.html